CLINICAL TRIAL: NCT03005613
Title: A Prospective, Randomized Comparison of Efficacy and Effect on Quality of Life Between Sacrospinous Ligament Fixation and Ischial Spine Fascia Fixation
Brief Title: Sacrospinous Ligament Fixation vs Ischial Spine Fascia Fixation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC-H0407-8160061244
Record Dates: First submitted 2016-12-15; First posted 2016-12-29 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2023-02

CONDITIONS: Urogenital Prolapse
Keywords: Pelvic organ prolapse; Sacrospinous ligament fixation; Ischial spine fascia fixation; Clinical outcome
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sacrospinous ligament fixation group (Active Comparator): The patients will receive sacrospinous ligament fixation operation.
  Interventions: Procedure: sacrospinous ligament fixation
- ischial spine fascia fixation group (Experimental): The patients will receive ischial spine fascia fixation operation.
  Interventions: Procedure: ischial spine fascia fixation

INTERVENTIONS:
Procedure: ischial spine fascia fixation — The participants will receive ischial spine fascia fixation.
  Arms: ischial spine fascia fixation group
Procedure: sacrospinous ligament fixation — The participants will receive sacrospinous ligament fixation.
  Arms: sacrospinous ligament fixation group

SUMMARY:
A Prospective, Randomized Comparison of Efficacy and Effect on Quality of Life Between Sacrospinous Ligament Fixation and Ischial Spine Fascia Fixation.

DETAILED DESCRIPTION:
Investigational intervention：SSLF or ISFF operations

Study title：A Prospective, Randomized Comparison of Efficacy and Effect on Quality of Life Between Sacrospinous Ligament Fixation and Ischial Spine Fascia Fixation.

Principal Investigator：Chang Ren, M.D., Department of Obstetrics & Gynecology, Peking Union Medical College Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College.

Study subjects：Adult patients with symptomatic stage II~IV pelvic organ prolapse will be eligible if all the inclusion criteria are met and without any reason for exclusion.

Study objectives：The primary objective of this study is to assess the short and mid-term efficacy of Sacrospinous Ligament Fixation and Ischial Spine Fascia Fixation in treating stage II~ IV pelvic organ prolapse and their recurrence rate as well as their impacts on quality of life.

Study design：Prospective, Single-Blind, Randomized, Clinical Trial

Intervention：

* ISFF group：Patients receive ISFF according to randomization.
* SSLF group：Patients receive SSLF according to randomization

Sample size：76 patients (38 in ISFF group, 38 in SSLF group)

Primary endpoint:

•objective success rates at 3 months after operations.

Secondary endpoints:

* peri-operative parameters .
* subjective satisfactory rates at 1 year after operations
* quality of life questionnaires at 1 year after operations

Safety endpoints: complications

ELIGIBILITY:
Inclusion Criteria:

* age≤65 years, for those scheduled to receive hysterectomy age≥40 years
* patients with symptomatic stage II~IV uterine or vaginal vault prolapse
* receiving SSLF or ISFF in the gynecological department at Peking Union Medical College Hospital

Exclusion Criteria:

* plans to live abroad within follow-up span
* contradiction to these two operations: acute genital infection, narrow vagina (less than two finger-breadth), too-ill to receive operations
* patients with hip joint problem who could not pose a lithotomy position

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
objective success | 3 months after operation
  no prolapse, stage I or only asymptomatic stage II prolapse

SECONDARY OUTCOMES:
Pelvic Floor Distress Inventory-20 (PFDI-20) | Change from Baseline in PFDI-20 at 3 months and 1 year
  to evaluate the quality of life in 3 domains
Pelvic Floor Impact Questionnaire-7 (PFIQ-7) | Change from Baseline in PFIQ-7 at 3 months and 1 year
  to evaluate the quality of life in 3 domains
Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire-12 (PISQ-12) | Change from Baseline in PISQ-12 at 3 months and 1 year
  to evaluate the sexual function
complications | through study completion, an average of 1 year
  peri-operative:massive bleeding, organ injury; post-operative: pelvic hematoma, pain, de novo UI, de novo dyspareunia
recurrence rate | 3 months after operation
  more than asymptomatic stage II prolapse after 3 months
subjective satisfaction ( according to a scale of 5 degrees: significantly worse, worse, no change, improved, greatly improved) | 1 year after operation
  Patient's response as improved or greatly improved

CONTACTS AND LOCATIONS:
Overall Officials: Chang Ren, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Department of Ob & Gyn, Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dwyer PL, Lee ET, Hay DM. Obesity and urinary incontinence in women. Br J Obstet Gynaecol. 1988 Jan;95(1):91-6. doi: 10.1111/j.1471-0528.1988.tb06486.x. PMID 3342213
- [Background] Sze EH, Karram MM. Transvaginal repair of vault prolapse: a review. Obstet Gynecol. 1997 Mar;89(3):466-75. doi: 10.1016/S0029-7844(96)00337-7. PMID 9052607
- [Background] Olsen AL, Smith VJ, Bergstrom JO, Colling JC, Clark AL. Epidemiology of surgically managed pelvic organ prolapse and urinary incontinence. Obstet Gynecol. 1997 Apr;89(4):501-6. doi: 10.1016/S0029-7844(97)00058-6. PMID 9083302
- [Background] Smith FJ, Holman CD, Moorin RE, Tsokos N. Lifetime risk of undergoing surgery for pelvic organ prolapse. Obstet Gynecol. 2010 Nov;116(5):1096-100. doi: 10.1097/AOG.0b013e3181f73729. PMID 20966694
- [Background] Boyles SH, Weber AM, Meyn L. Procedures for pelvic organ prolapse in the United States, 1979-1997. Am J Obstet Gynecol. 2003 Jan;188(1):108-15. doi: 10.1067/mob.2003.101. PMID 12548203
- [Background] Barber MD, Maher C. Apical prolapse. Int Urogynecol J. 2013 Nov;24(11):1815-33. doi: 10.1007/s00192-013-2172-1. PMID 24142057
- [Background] Jones KA, Shepherd JP, Oliphant SS, Wang L, Bunker CH, Lowder JL. Trends in inpatient prolapse procedures in the United States, 1979-2006. Am J Obstet Gynecol. 2010 May;202(5):501.e1-7. doi: 10.1016/j.ajog.2010.01.017. Epub 2010 Mar 11. PMID 20223444
- [Background] Zhu L, Lang J, Zhang Q. Clinical study of ischia spinous fascia fixation--a new pelvic reconstructive surgery. Int Urogynecol J. 2011 Apr;22(4):499-503. doi: 10.1007/s00192-010-1307-x. PMID 21060988